CLINICAL TRIAL: NCT02485288
Title: PaTH Clinical Data Research Network (CDRN) Atrial Fibrillation (AF) Clinician-Patient Partnership Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Johns Hopkins University (Other); Penn State University (Other); Temple University (Other)
Responsible Party: Principal Investigator, Kathleen McTigue, Professor, University of Pittsburgh
Other Study IDs: STUDY20110294
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the PaTH Network AF Clinician-Patient Partnership Cohort is to use clinical data from electronic health records (EHR) and patient reported outcomes (PRO) to answer questions of clinical importance to patients, providers, and other stakeholders.

DETAILED DESCRIPTION:
The primary objective is to create the PaTH Network AF Clinician-Patient Partnership Cohort, which will allow the conduct of patient-centered observational studies on AF across the multiple institutions of the PaTH network. Creating the AF Clinician-Patient Partnership Cohort will involve:

1. Recruiting patients with AF to participate in the PaTH Network AF Clinician-Patient Partnership Cohort
2. Administering surveys to the AF Clinician-Patient Partnership Cohort approximately every 6 months to collect patient reported outcomes (PROs)
3. Collecting individual patient health record data into the AF Clinician-Patient Partnership Cohort database
4. Tracking whether the patient participant has biospecimens in a PaTH site biorepository and prepare for possible sharing of biospecimens in future studies.
5. Identifying potential participants for future research studies.

The secondary objectives are to use the PaTH Network AF Clinician-Patient Partnership Cohort to answer patient-centered research questions including:

1. What is the incidence of complications requiring re-hospitalization after an ablation procedure for AF?
2. What are the predictors of major bleeding and stroke among patients that receive each anticoagulant class (vit K antagonist, direct factor X inhibitor, direct thrombin inhibitor)?
3. Is the longitudinal change in applied cognition-executive function score in AF patients associated with the choice of rate versus rhythm control and anticoagulation strategy?

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older at time of query
* Visits: 3 non-ED outpatient visits between 1/1/2011 and 12/31/2014
* AF : AF diagnosis documented between 1/1/2011 and 12/31/2014
* AF diagnosis can be coded EHR (on billing or problem lists) and/or derived from EKG reports
* AF diagnoses associated with surgery, certain thyroid conditions, or certain medications cannot count as the qualifying AF diagnosis for inclusion in this cohort.

Exclusion Criteria:

* Deceased
* Not proficient in English
* Already enrolled in the PaTH Clinical Data Research Network (CDRN) Atrial Fibrillation (AF) Clinician-Patient Partnership Cohort at another PaTH institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants for the PaTH Clinical Data Research Network (CDRN) Atrial Fibrillation (AF) Clinician-Patient Partnership Cohort will include patients identified through EHRs at the participating PaTH sites, using the eligibility criteria described below. We aim to recruit as many patients as possible from the target population, with one of the recruitment strategies producing a 50% enrollment rate.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-06; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Create PaTH Clinical Data Research Network (CDRN) Atrial Fibrillation (AF) Clinician-Patient Partnership Cohort | 18 months
  Create the PaTH Clinical Data Research Network (CDRN) Atrial Fibrillation (AF) Clinician-Patient Partnership Cohort which will allow the conduct of patient-centered observational studies on atrial fibrillation across the multiple institutions (Hershey Penn State, University of Pittsburgh, Temple University) of the PaTH network.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M McTigue, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Jody McCullough, Hershey, Pennsylvania
  - Anuradha Paranjape, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Gleason KT, Dennison Himmelfarb CR, Ford DE, Lehmann H, Samuel L, Han HR, Jain SK, Naccarelli GV, Aggarwal V, Nazarian S. Association of sex, age and education level with patient reported outcomes in atrial fibrillation. BMC Cardiovasc Disord. 2019 Apr 5;19(1):85. doi: 10.1186/s12872-019-1059-6. PMID 30953478
- [Background] Gleason KT, Dennison Himmelfarb CR, Ford DE, Lehmann H, Samuel L, Jain S, Naccarelli G, Aggarwal V, Nazarian S. Association of sex and atrial fibrillation therapies with patient-reported outcomes. Heart. 2019 Nov;105(21):1642-1648. doi: 10.1136/heartjnl-2019-314881. Epub 2019 May 22. PMID 31118198